CLINICAL TRIAL: NCT03421834
Title: Impact of PREVENTIVE Substrate Catheter Ablation on Implantable cardioVerter-defibrillaTor Interventions in Patients With Ischaemic Cardiomyopathy and Infarct-related Coronary Chronic Total Occlusion
Brief Title: Impact of PREVENTIVE Substrate Ablation of Coronary Chronic Total Occlusion on Implantable cardioVerTer-Defibrillator Interventions
Acronym: PREVENTIVE VT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, David Žižek, MD, PhD, Assistant Professor, Principal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREVENTIVE VT
Record Dates: First submitted 2018-01-25; First posted 2018-02-05 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Ventricular Tachycardia; Ischemic Cardiomyopathy
Keywords: Ventricular Tachycardia; Ischemic Cardiomyopathy; Primary prevention; Heart Failure
MeSH Terms: conditions — Tachycardia, Ventricular; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic VT ablation prior to ICD implantation (Experimental)
  Interventions: Procedure: Catheter ablation of ventricular tachycardia; Drug: Optimal medical treatment
- ICD implantation and optimal medical treatment (Active Comparator): ICD implantation and optimal medical care until at least 2 appropriate ICD shock occurs or an arrhythmic storm and catheter ablation thereafter.
  Interventions: Drug: Optimal medical treatment

INTERVENTIONS:
Procedure: Catheter ablation of ventricular tachycardia — Catheter ablation with a uniform mapping system, procedural endpoint, and definition of acute procedural success.
  Arms: Prophylactic VT ablation prior to ICD implantation
Drug: Optimal medical treatment — Optimal guidelines-based heart failure treatment and antiarrhythmic drugs. Antiarrhythmics will be avoided if possible in the ablation group.

SUMMARY:
The aim of this study is to assess whether preventive substrate ablation of chronic total occlusion infarct-related artery (CTO-IRA) area in heart failure (HF) patients correlates with lower appropriate implantable cardiac defibrillator (ICD) therapies. In addition, the purpose of the study is to determine whether prophylactic substrate ablation at the time of primary ICD implantation in high-risk ischemic patients affects unplanned hospitalization, HF progression, and quality of life.

DETAILED DESCRIPTION:
Implantable cardioverter-defibrillators (ICDs) improve survival among patients with ischemic heart failure (HF) who have not previously had a sustained ventricular arrhythmia. However, ICD shocks that terminate ventricular tachycardia (VT) are associated with higher mortality, which may be a reflection of ICD shocks being a marker of more advanced disease versus shocks causing a worse prognosis. In addition, ICD shocks are associated with decreased functional status and quality of life. Antiarrhythmic medications (AAD) reduce ICD shocks but have high rates of side effects and lack of compliance within 1 year of initiation. Some randomized, controlled clinical trials have shown that catheter ablation (CA) of VT can decrease the number of episodes of VT and ICD shocks which could translate to an improvement in patient outcomes.

Regarding the approach to CA of VT, several controversies and gaps of knowledge can be found in the literature. Some authors target predominantly "clinical VTs" (activation and entrainment mapping), while others focus on the substrate causing VTs without focusing on VT morphologies (elimination of local abnormal ventricular activities and late potentials). In addition, data on timing of the CA procedure is inconsistent. However, early CA strategy seems feasible as end-stage cardiovascular disease increases procedural risk and is associated with arrhythmias that may be less amenable to successful treatment with ablation.

The current focus on risk stratifying patients with ischemic cardiomyopathy who could benefit from a primary prevention ICD solely on basis of ejection fraction and NYHA class is far from ideal. In patients with ischemic HF, the presence of the coronary chronic total occlusion (CTO) is related to worse long-term prognosis. Moreover, in a subgroup of ischemic patients, CTO associated with a previous infarction in its territory was an independent predictor of ventricular arrhythmias. Recent studies reported that primary prevention patients with CTO of an infarct-related artery (CTO-IRA) have a very high risk of appropriate ICD therapies due to fast VTs. As post-myocardial infarction scar is a well-recognized substrate of VTs, these patients might benefit from prophylactic substrate ablation at the time of primary ICD implantation.

Eligible and consenting patients on optimal medical HF treatment with confirmed CTO-IRA will be equally randomized to receive either a primary prevention ICD or a CA procedure and an ICD. Catheter ablation with a uniform procedural endpoint and definition of acute procedural success was to be performed before ICD implantation. ICD programming will be standardized for all subjects according to primary prevention settings.

Subjects will be seen at baseline randomization, then 1 month after ICD implantation and every 6 months thereafter until the end of the study. Subjects will be followed up for a minimum of 24 months. Quality of life questionnaires will be done at each visit.

The aim of this study is to assess whether preventive substrate ablation of CTO-IRA area in HF patients correlates with lower appropriate ICD therapies. In addition, the purpose of the study is to determine whether prophylactic substrate ablation at the time of primary ICD implantation in high-risk ischemic patients affects unplanned hospitalization, HF progression, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic cardiomyopathy with reduced ejection fraction (EF ≤ 40%) estimated by cardiac MRI or echocardiography within 30 days before enrollment
2. Coronary Chronic Total Occlusion (CTO) associated with a previous MI confirmed by coronary angiography and late gadolinium enhancement MRI or myocardial perfusion imaging within 30 days before enrollment
3. Implantable cardioverter-defibrillator (ICD) indication for primary prevention
4. Patient has provided written informed consent

Exclusion Criteria:

1. Age < 18 years or > 85 years
2. Documented sustained ventricular tachycardia before enrollment
3. Class IV New York Heart Association (NYHA) heart failure
4. CTOs not associated with a prior infarction in their territory
5. Acute myocardial infarction (MI) or acute coronary syndrome
6. Subjects with active ischemia that are eligible for revascularization
7. Documented history of MI less than 6 months before enrollment
8. Patients requiring chronic renal dialysis
9. Thrombocytopenia or coagulopathy
10. Pre-existing implantable cardioverter-defibrillator (ICD)
11. Pregnancy or breastfeeding women
12. Acute illness or active systemic infection
13. Life expectancy less than 12 months
14. Unwillingness to participate or lack of availability for follow-up
15. Valvular heart disease or mechanical heart valve precluding access to the left ventricle

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Time to first event comprising appropriate ICD therapy and unplanned hospital admission for symptomatic ventricular tachycardia (VT)/ ventricular fibrillation (VF) | From randomization until official study end or drop-out, patients will be followed and assessed at least 24 months.
  Appropriate ICD therapy defined as shock or ATP therapy.

SECONDARY OUTCOMES:
Time to appropriate ICD therapy | At least 24 months after enrolment
  Appropriate ICD therapy defined as shock or ATP therapy.
Incidence of appropriate ICD therapy | At least 24 months after enrolment
Time to unplanned hospital admission for symptomatic ventricular tachycardia (VT)/ ventricular fibrillation (VF) | At least 24 months after enrolment
Time to unplanned cardiac hospital admission | At least 24 months after enrolment
Time to electrical storm | At least 24 months after enrolment
  Electrical storm defined by 3 or more sustained episodes of ventricular tachycardia (VT), ventricular fibrillation (VF), or appropriate ICD therapy within 24 hours.
Cardio-vascular mortality | At least 24 months after enrolment
Changes in quality of life using the EQ-5D questionnaire | At least 24 months after enrolment
  EQ-5D is a standardised measure of health status consisting of 2 pages - the EQ-5D descriptive system (descriptive system with 3 levels) and the EQ visual analogue scale ranging from 0 (worst state) to 100 (best state).
Psychometric evaluation of ICD shock-related anxiety using The Florida Shock Anxiety Scale (FSAS) | At least 24 months after enrolment
  Questions were designed to capture patient opinion on perceptions of current health status, as well as a subjective opinion of how the ICD has affected them in specific areas, including anxiety levels. A higher score indicates an positive response and a lower score indicates a negative response.

CONTACTS AND LOCATIONS:
Overall Officials: Matjaz Sinkovec, Prof., Study Chair — University Medical Centre Ljubljana (Slovenia); Andrej Pernat, Prof., Study Chair — University Medical Centre Ljubljana (Slovenia); David Zizek, Assist. Prof., Principal Investigator — University Medical Centre Ljubljana (Slovenia)
Locations (5):
- Klinički bolnički centar Sestre Milosrdnice, Zagreb, Croatia
- Slovenia (4):
  - General Hospital Celje, Celje
  - General Hospital Izola, Izola
  - University Medical Centre Ljubljana - Cardiology department, Ljubljana
  - University Medical Centre Ljubljana - Cardiovascular surgery department, Ljubljana

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Poole JE, Johnson GW, Hellkamp AS, Anderson J, Callans DJ, Raitt MH, Reddy RK, Marchlinski FE, Yee R, Guarnieri T, Talajic M, Wilber DJ, Fishbein DP, Packer DL, Mark DB, Lee KL, Bardy GH. Prognostic importance of defibrillator shocks in patients with heart failure. N Engl J Med. 2008 Sep 4;359(10):1009-17. doi: 10.1056/NEJMoa071098. PMID 18768944
- [Background] Reddy VY, Reynolds MR, Neuzil P, Richardson AW, Taborsky M, Jongnarangsin K, Kralovec S, Sediva L, Ruskin JN, Josephson ME. Prophylactic catheter ablation for the prevention of defibrillator therapy. N Engl J Med. 2007 Dec 27;357(26):2657-65. doi: 10.1056/NEJMoa065457. PMID 18160685
- [Background] Dinov B, Arya A, Bertagnolli L, Schirripa V, Schoene K, Sommer P, Bollmann A, Rolf S, Hindricks G. Early referral for ablation of scar-related ventricular tachycardia is associated with improved acute and long-term outcomes: results from the Heart Center of Leipzig ventricular tachycardia registry. Circ Arrhythm Electrophysiol. 2014 Dec;7(6):1144-51. doi: 10.1161/CIRCEP.114.001953. Epub 2014 Sep 27. PMID 25262159
- [Background] Di Biase L, Burkhardt JD, Lakkireddy D, Carbucicchio C, Mohanty S, Mohanty P, Trivedi C, Santangeli P, Bai R, Forleo G, Horton R, Bailey S, Sanchez J, Al-Ahmad A, Hranitzky P, Gallinghouse GJ, Pelargonio G, Hongo RH, Beheiry S, Hao SC, Reddy M, Rossillo A, Themistoclakis S, Dello Russo A, Casella M, Tondo C, Natale A. Ablation of Stable VTs Versus Substrate Ablation in Ischemic Cardiomyopathy: The VISTA Randomized Multicenter Trial. J Am Coll Cardiol. 2015 Dec 29;66(25):2872-2882. doi: 10.1016/j.jacc.2015.10.026. PMID 26718674
- [Background] Nombela-Franco L, Mitroi CD, Fernandez-Lozano I, Garcia-Touchard A, Toquero J, Castro-Urda V, Fernandez-Diaz JA, Perez-Pereira E, Beltran-Correas P, Segovia J, Werner GS, Javier G, Luis AP. Ventricular arrhythmias among implantable cardioverter-defibrillator recipients for primary prevention: impact of chronic total coronary occlusion (VACTO Primary Study). Circ Arrhythm Electrophysiol. 2012 Feb;5(1):147-54. doi: 10.1161/CIRCEP.111.968008. Epub 2011 Dec 28. PMID 22205684
- [Background] Di Marco A, Anguera I, Teruel L, Dallaglio P, Gonzalez-Costello J, Leon V, Nunez E, Manito N, Gomez-Hospital JA, Sabate X, Cequier A. Chronic total occlusion of an infarct-related artery: a new predictor of ventricular arrhythmias in primary prevention implantable cardioverter defibrillator patients. Europace. 2017 Feb 1;19(2):267-274. doi: 10.1093/europace/euw009. PMID 28175266
- [Background] Di Marco A, Anguera I, Teruel L, Muntane G, Campbell NG, Fox DJ, Brown B, Skene C, Davidson N, Leon V, Dallaglio P, Elzein H, Garcia-Romero E, Gomez-Hospital JA, Cequier A. Chronic total occlusion in an infarct-related coronary artery and the risk of appropriate ICD therapies. J Cardiovasc Electrophysiol. 2017 Oct;28(10):1169-1178. doi: 10.1111/jce.13290. Epub 2017 Aug 4. PMID 28675508
- [Derived] Kheiri B, Barbarawi M, Zayed Y, Hicks M, Osman M, Rashdan L, Kyi HH, Bachuwa G, Hassan M, Stecker EC, Nazer B, Bhatt DL. Antiarrhythmic Drugs or Catheter Ablation in the Management of Ventricular Tachyarrhythmias in Patients With Implantable Cardioverter-Defibrillators: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Circ Arrhythm Electrophysiol. 2019 Nov;12(11):e007600. doi: 10.1161/CIRCEP.119.007600. Epub 2019 Nov 8. PMID 31698933